CLINICAL TRIAL: NCT03775603
Title: Comparison of TOFscan and TOF-Watch SX in Children
Brief Title: Comparison of TOFscan and TOF-Watch SX in Pediatric Neuromuscular Function Recovery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, principal investigator, Seoul National University Hospital
Other Study IDs: 1811-137-989
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TOFscan — comparison of TOFscan over TOF-Watch SX

SUMMARY:
Comparison of TOFscan and TOF-Watch SX for monitoring of neuromuscular blockade function in children

DETAILED DESCRIPTION:
TOF ratio of TOFscan when TOF-Watch SX shows TOF ratio 0.7 with rocuronium in children during general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* patients need neuromuscular blockade

Exclusion Criteria:

* contraindication of rocuronium

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: general anesthesia with neuromuscular blockade in children
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
TOF ratio of TOFscan | intraoperative during anesthesia
  value of TOF ratio of TOFscan at TOF ratio 0.7 of TOF-Watch SX during neuromuscular function recovery period

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yhim HB, Jang YE, Lee JH, Kim EH, Kim JT, Kim HS. Comparison of the TOFscan and the TOF-Watch SX during pediatric neuromuscular function recovery: a prospective observational study. Perioper Med (Lond). 2021 Dec 10;10(1):45. doi: 10.1186/s13741-021-00215-2. PMID 34886885